CLINICAL TRIAL: NCT03516422
Title: Ultrasound Debridement In Chronic Lower Extremity Wounds - A Pilot Study
Brief Title: Investigating Ultrasound Debridement in Wound Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16-187
Record Dates: First submitted 2016-07-29; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Diabetes
Keywords: ultrasound debridement; diabetic foot ulcer; chronic wound; biofilm
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STANDARD CARE GROUP (Placebo Comparator): The subject positioned so absorbent pads are in position to catch irrigation solution. The saline bottle will be held 10-15 cm from wound bed, and squeezed to spray all surfaces of wound in a sweeping motion, from clean to dirty area of wound. Irrigation will be repeated as necessary to remove exudate, slough, and debris from the wound until the solution draining from the wound is clear. Peri-wound skin will be cleansed using gauze and sterile normal saline and dry. Packing material will be applied (Acticoat®) into the wound cavity, undermining, or tunnel to fill the dead space without causing the wound to stretch or bulge or be packed tightly. Packing should be in contact with entire wound base and edges. Dressings changed once every 3 days by the patient's care provider.
  Interventions: Other: STANDARD CARE GROUP
- ULTRASOUND DEBRIDEMENT GROUP: (Experimental): Low-frequency ultrasound SonicOne O.R. (Misonix, New York, US) generates ultrasound waves with 22.5 kHz frequency. Each probe is attached to a set of irrigation solution (saline 0.9%), they transform electric energy into mechanical vibrations to induce tiny particles of water from irrigation fluid. Absorbent pads are positioned to catch excess saline. With SonicOne set at continuous mode with minimum pump flow, the debridement will begin at most distal aspect of ulcer with the hand piece in constant motion until entire ulcer surface has been debrided until as much necrotic tissue has been removed. Peri-wound skin will be cleansed using gauze and sterile normal saline and dry. Packing material will be applied (Acticoat®) into wound cavity.
  Interventions: Procedure: ULTRASOUND DEBRIDEMENT

INTERVENTIONS:
Procedure: ULTRASOUND DEBRIDEMENT — Low-frequency ultrasound SonicOne O.R. (Misonix, New York, US) generates ultrasound waves with 22.5 kHz frequency. Each probe is attached to a set of irrigation solution (saline 0.9%), they transform electric energy into mechanical vibrations to induce tiny particles of water from irrigation fluid. Absorbent pads are positioned to catch excess saline. With SonicOne set at continuous mode with minimum pump flow, the debridement will begin at most distal aspect of ulcer with the hand piece in constant motion until entire ulcer surface has been debrided until as much necrotic tissue has been removed. Peri-wound skin will be cleansed using gauze and sterile normal saline and dry. Packing material will be applied (Acticoat®) into wound cavity.
  Arms: ULTRASOUND DEBRIDEMENT GROUP:
Other: STANDARD CARE GROUP — The subject positioned so absorbent pads are in position to catch irrigation solution. The saline bottle will be held 10-15 cm from wound bed, and squeezed to spray all surfaces of wound in a sweeping motion, from clean to dirty area of wound. Irrigation will be repeated as necessary to remove exudate, slough, and debris from the wound until the solution draining from the wound is clear. Peri-wound skin will be cleansed using gauze and sterile normal saline and dry. Packing material will be applied (Acticoat®) into the wound cavity, undermining, or tunnel to fill the dead space without causing the wound to stretch or bulge or be packed tightly. Packing should be in contact with entire wound base and edges. Dressings changed once every 3 days by the patient's care provider.
  Arms: STANDARD CARE GROUP

SUMMARY:
The initial step of wound management, debridement, is thought to be critical in promoting wound healing. Of the numerous debridement modalities, ultrasound seems to hold promising results in accelerate healing in our own clinical experience here at St. Michael's Hospital. In brief, ultrasound debridement is a method of removing devitalized tissue through microstreaming and cavitational effects. The non-thermal energy up-regulates cellular activity and promotes growth factor and protein synthesis, fibrinolysis, and is anti-bacterial . The technology selectively emulsifies dead and dying tissues with micro-sized gas bubbles, stimulates membranes of surrounding healthy cells, and renders bacteria more susceptible to antibiotic treatment. Thus, in addition to creating an optimal environment, the modality also serves to promote the process of healing. A systematic review and meta-analysis by Voigt et al. (2011) examined the use of low-frequency (20-30 kHz) ultrasound in randomized-controlled trials. It was found that low or high-intensity delivery of low-frequency ultrasound both promoted early healing in lower-extremity wounds. At St. Michael's Hospital, ultrasound debridement is already being used in the wound clinic with promising results. However, objective comparisons need to be made to validate our clinical observations. The goal of the proposed pilot study is to assess the feasibility of our current study design. The information gathered will allow us to refine the research methodology for the development of a larger-scale study.

DETAILED DESCRIPTION:
Ultrasound debridement is a method of removing devitalized tissue through microstreaming and cavitational effects. The non-thermal energy up-regulates cell activity and promotes growth factor and protein synthesis, fibrinolysis, and is anti-bacterial. The technology selectively emulsifies dead and dying tissues with micro-sized gas bubbles, stimulates membranes of surrounding healthy cells, and render bacteria more susceptible to antibiotic treatment. Thus, in addition to creating an optimal environment, the modality also serves to promote the process of healing. At St. Michael's Hospital, ultrasound debridement is already being used in the wound clinic with promising results. However, objective comparisons need to be made to quantify and qualify our clinical observations. The goal of the proposed pilot study is to assess feasibility of our current study design and allow us to refine the research methodology for the development of a larger-scale study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with chronic (>4 week duration) lower extremity wound (of any etiology) that have failed to improve despite using the clinic's standard approach for wound care during a 2-week period (Failure to improve is defined as less than 15% reduction in wound area)

Exclusion Criteria:

1. Subjects with clinical evidence of wound infection
2. Subjects with thick eschar that has not been removed
3. Subjects with severe arterial insufficiency: Absence of pedal pulses, Ankle Brachial Index < 0.3, Toe Pressure < 20
4. Subjects who are receiving advanced wound therapy treatment: hyperbaric therapy, biological dressings
5. Subjects who are taking antibiotics
6. Subjects who are using systemic steroids
7. Subjects who have known contraindication to the dressing product (Acticoat®)
8. Subjects who are not able to adhere to dressing change protocol or hospital visits
9. Subjects with wound area reduction of > 15% during the initial two-week standard care period.
10. Subjects without sufficient English language proficiency to understand the consent form.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Wound healing | 8 weeks
  Healing of the wound

SECONDARY OUTCOMES:
Change in biofilm microbiome | 8 weeks
  Shift in biofilm to reflect wound healing
Reduction in bacterial colonization | 8 weeks
  Decreased bacterial colonization to reflect wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cross, MD, PhD, Principal Investigator — Staff Plastic Surgeon

IPD SHARING:
Plan to Share IPD: No
No sharing of data

REFERENCES:
- [Background] Alguire PC, Mathes BM. Skin biopsy techniques for the internist. J Gen Intern Med. 1998 Jan;13(1):46-54. doi: 10.1046/j.1525-1497.1998.00009.x. PMID 9462495
- [Background] Altland OD, Dalecki D, Suchkova VN, Francis CW. Low-intensity ultrasound increases endothelial cell nitric oxide synthase activity and nitric oxide synthesis. J Thromb Haemost. 2004 Apr;2(4):637-43. doi: 10.1111/j.1538-7836.2004.00655.x. PMID 15102020
- [Background] Gardner SE, Frantz RA, Saltzman CL, Hillis SL, Park H, Scherubel M. Diagnostic validity of three swab techniques for identifying chronic wound infection. Wound Repair Regen. 2006 Sep-Oct;14(5):548-57. doi: 10.1111/j.1743-6109.2006.00162.x. PMID 17014666
- [Background] Miller CN, Newall N, Kapp SE, Lewin G, Karimi L, Carville K, Gliddon T, Santamaria NM. A randomized-controlled trial comparing cadexomer iodine and nanocrystalline silver on the healing of leg ulcers. Wound Repair Regen. 2010 Jul-Aug;18(4):359-67. doi: 10.1111/j.1524-475X.2010.00603.x. PMID 20636550
- [Background] Sibbald RG, Woo K, Ayello EA. Increased bacterial burden and infection: the story of NERDS and STONES. Adv Skin Wound Care. 2006 Oct;19(8):447-61; quiz 461-3. doi: 10.1097/00129334-200610000-00012. PMID 17008815
- [Background] Wu YC, Kulbatski I, Medeiros PJ, Maeda A, Bu J, Xu L, Chen Y, DaCosta RS. Autofluorescence imaging device for real-time detection and tracking of pathogenic bacteria in a mouse skin wound model: preclinical feasibility studies. J Biomed Opt. 2014 Aug;19(8):085002. doi: 10.1117/1.JBO.19.8.085002. PMID 25089944